CLINICAL TRIAL: NCT01004926
Title: Evaluation of the Efficiency of the Echelon Foot in Traumatic Trans Tibial
Brief Title: Evaluation of the Efficiency of the Echelon Foot in Traumatic Trans Tibial Amputees
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Itzhak Siev-Ner, Dr. Itzhak Siev-Ner, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-09-7325-IS-CTIL
Record Dates: First submitted 2009-10-19; First posted 2009-10-30 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Unilateral Trans Tibial Amputation
Keywords: Unilateral trans-tibial amputees

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Echelon (Experimental)
  Interventions: Device: Echelon foot

INTERVENTIONS:
Device: Echelon foot — One Echelon foot for each subject, for a period of a month.

SUMMARY:
The aim of this work was to test the Echelon foot efficiency to offer enhanced safety, comfort and function over a wide range of walking surfaces, inclines and stairs, thereby improving the quality of life for amputees.

Ten individuals with a unilateral trans- tibial amputation will participate in two test sessions- one while using their own prosthetic foot, the other while using the Echelon foot.

ELIGIBILITY:
Inclusion Criteria:

* Ten individuals with a unilateral trans tibial amputation due to trauma.
* Walking at list one year from the end of their gait training. Mobility status is 3 or 4.

Exclusion Criteria:

* Bilateral amputation.
* Injury of the sound limb that compromises the gait of the amputee.

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
While using the Echelon foot the amputees will present lower internal mechanical strain in the soft tissue of the stump while standing on a 10 degrees platform. | Beginning of the trial and one month after

SECONDARY OUTCOMES:
Using the Echelon foot the Kinematic of level ground walking and climbing up and down stairs will be closer to normal curves. | At the beginning of the trial and one month later

CONTACTS AND LOCATIONS:
Overall Officials: Itzhak Siev- Ner, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel